CLINICAL TRIAL: NCT00091429
Title: A Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Study of Ranolazine SR at a Dose of 1000 mg Twice a Day in Patients With Chronic Angina Who Remain Symptomatic Despite Treatment With Amlodipine 10 mg Once a Day
Brief Title: Ranolazine SR in Patients With Chronic Angina Who Remain Symptomatic Despite Maximal Treatment With Amlodipine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Philip Sager, Vice President, Clinical Research, Gilead Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVT 3037
Record Dates: First submitted 2004-09-08; First posted 2004-09-10 (Estimated); Last update posted 2009-11-26 (Estimated); Status verified 2009-11

CONDITIONS: Angina
Keywords: Angina; Chest Pain; Coronary Artery Disease; Heart Disease
MeSH Terms: conditions — Angina Pectoris; Chest Pain; Coronary Artery Disease; Heart Diseases | interventions — Ranolazine

INTERVENTIONS:
Drug: Ranolazine

SUMMARY:
The study will be a multi-national, double-blind, randomized, placebo-controlled, parallel group study to evaluate the effectiveness of ranolazine (1000 mg twice daily) in approximately 500 patients with chronic angina who remain symptomatic despite daily treatment with the maximum labeled dose of amlodipine (10 mg daily), a calcium channel blocker approved for the treatment of chronic angina. Eligible patients will be randomized to receive ranolazine 1000 mg or placebo twice daily, in addition to a daily dose of 10 mg of amlodipine. Participation in the study will last approximately 3 months.

ELIGIBILITY:
Eligible patients must have a diagnosis of chronic angina, with documented evidence of coronary artery disease or prior myocardial infarction, in addition to other study entry criteria. Prior to entering the study, patients will be required to have had at least two weeks of treatment with amlodipine 10 mg daily, with the discontinuation of all other anti-anginal therapy for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2004-08; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

REFERENCES:
- [Result] Stone PH, Gratsiansky NA, Blokhin A, Huang IZ, Meng L; ERICA Investigators. Antianginal efficacy of ranolazine when added to treatment with amlodipine: the ERICA (Efficacy of Ranolazine in Chronic Angina) trial. J Am Coll Cardiol. 2006 Aug 1;48(3):566-75. doi: 10.1016/j.jacc.2006.05.044. Epub 2006 Jun 15. PMID 16875985
- [Derived] Kohn CG, Parker MW, Limone BL, Coleman CI. Impact of angina frequency on health utility values of patients with chronic stable angina. Health Qual Life Outcomes. 2014 Mar 14;12:39. doi: 10.1186/1477-7525-12-39. PMID 24628859